CLINICAL TRIAL: NCT01661985
Title: Study of Time to Eradication of Mycoplasma Genitalium and Chlamydia Trachomatis After Antibiotic Treatment
Brief Title: Time to Eradication of Mycoplasma Genitalium and Chlamydia Trachomatis After Treatment Commenced
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Lars Falk, MD PhD, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ostergotland CC
Record Dates: First submitted 2012-07-27; First posted 2012-08-10 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Urethritis; Cervicitis; Genital Mycoplasma Infection; Chlamydia Trachomatis
Keywords: Mycoplasma genitalium; Chlamydia trachomatis; Treatment; Antibiotic resistance
MeSH Terms: conditions — Urethritis; Uterine Cervicitis | interventions — Azithromycin; Doxycycline; Lymecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Drug: Azithromycin 1g (Active Comparator): Azithromycin 1 g,single dose (per os)
  Interventions: Drug: Azithromycin
- Drug: Doxycycline/lymecycline 9/10days (Active Comparator): Tetracycline either as Doxycycline or during June and July lymecycline (due to lower risk of photo-sensitivity) given for treatment in 9(10)days (per os).
  Interventions: Drug: Doxycycline; Drug: lymecycline
- Azithromycin 1.5 g (Active Comparator): Patients not randomized but receiving the first line treatment when a confirmed Mg infection
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — In the randomized arm giver orally 1 g as a single dose. In the non-randomized arm given for 5 days 250mg 2x1 first day and 1x1 following four days.
  Other Names: Zitromax; Azitromax
  Arms: Azithromycin 1.5 g; Drug: Azithromycin 1g
Drug: Doxycycline — Doxycycline tablets 100 mg 2x1 the first day and 100 mg daily for following eight days (following the Swedish tradition and experience since the 1970s of treating chlamydia)
  Other Names: Doxyferm
  Arms: Drug: Doxycycline/lymecycline 9/10days
Drug: lymecycline — Lymecycline 300 mg twice daily for 10 days (Summertime due to less risk of phototoxic reactions)
  Other Names: Tetralysal 300mg
  Arms: Drug: Doxycycline/lymecycline 9/10days

SUMMARY:
The purpose of this on-going study is to study the number of days after antibiotic treatment has commenced (due to infection caused by the sexually transmitted bacteria Chlamydia trachomatis (CT) and Mycoplasma genitalium(Mg)) it takes to be cured i.e to get a negative test result. The specimens are analyzed on first-catch-urine (men) or patient's self-obtained vaginal sample with quantitive nucleic acid amplification test(NAAT). A secondary aim is to detect macrolide resistant Mg-strains and study whether there are any emerging macrolide resistant Mg-strains after treatment with azithromycin. A third aim is to study whether the participating subjects are adherent to the study protocol meaning 12 samples taken during a period of four weeks.

DETAILED DESCRIPTION:
Mycoplasma genitalium (Mg), detected in 1980, causes a urogenital infection through sexual transmission. In contrast to Chlamydia trachomatis antibiotic resistance is common against tetracyclines and is emerging against macrolides such as azithromycin. Both antibiotics are recommended as the first line treatment of chlamydia infection. Recent published data, however, indicate that 1g azithromycin stat may be only bacteriostatic when treating chlamydia.

The consensus to date is that there should always be a test of cure in pregnant women having been treated for chlamydia and in all individuals treated for Mg.

There are no studies published, to our knowledge, where the time to eradication after antibiotic treatment commenced in Mg infection has been evaluated. The first line treatment of a confirmed Mg infection is azithromycin 1.5 g given during a period of 5 days. If macrolide resistance is plausible or confirmed moxifloxacin 400mg for 7 to 10 days is recommended.

Individuals with symptomatic urethritis or cervicitis and/or being sexual partners to individuals being treated for a suspect or confirmed Mg or CT infection were eligible. The study subjects were patients attending either of the STD-clinics in Norrköping or Västervik, Sweden. All samples were sent to Statens Serum Institut(SSI), Mycoplasma department (Jorgen Skov Jensen) for analysis.

Patients accepting enrolment with a confirmed or highly suspected Mg were receiving azithromycin 500 mg the first day and 250mg the following four days.

Patients where macrolide resistant Mg-strain infection was highly suspected received moxifloxacin 400 mg once daily for seven days.

Those subjects intended to treatment but with a lower degree of suspicion of Mg infection were randomized to either a treatment with doxycycline 200 mg the first day and 100 mg once daily the following nine days (the custom and recommendation in Sweden for treatment of chlamydia and non-specific urethritis or cervicitis) OR a treatment with azithromycin 1g as a single dose.

All participants were given test kits for 12 samples, which were to be sampled three times weekly (every second day) during four weeks starting the day after the first day of treatment. They were instructed not to have any sexual intercourse during the first week and with condom afterwards during the study period. The samples were to be sent once weekly (three samples)to SSI.The date of sampling was to be noted on the label of the tube and the attaching paper to SSI, where also any symptoms were to be noted. The results of the tests were sent to the STD-clinic who informed the patient.

The study started in February 2010 and inclusion of patients have ended for those subjects with a verified M genitalium infection (February 2014), whereas patients with a verified or suspected chlamydia infection still are enrolled and randomised to azithromycin 1 g or doxycycline. A manuscript will soon be submitted concerning those subjects being treated for a M genitalium infection.

To date 190 patients have been enrolled and also fulfilled the study protocol with sampling of specimens.

ELIGIBILITY:
Inclusion Criteria:

* Individuals attending the STD-clinic and being a sexual partner who has received an antibiotic treatment due to a non-specific urethritis/cervicitis or a confirmed Mycoplasma genitalium/Chlamydia trachomatis infection OR Having a confirmed infection described above or a symptomatic urethritis or cervicitis (non-gonorrhoic)

Exclusion Criteria:

* Allergy against any of the drugs, woman being pregnant or breast feeding, Not speaking or understanding Swedish fluently. Other medication with possible interaction to given treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-02; Primary Completion 2015-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Time from treatment starts to date of first negative test result is achieved up to 30 days. | From first day of treatment to date of first negative test up to 30 days per subject
  Three arms. A randomisation (concealed envelopes) to either treatment with azithromycin 1g as a single dose or doxycycline for nine days (200 mg first day and 100 mg following nine (during summer time lymecycline 300mg twice daily for ten days). One un-randomized arm: Treatment with azithromycin 500 mg the first day and 250mg following four days or when indicated moxifloxacin 400 mg once daily for seven days.

SECONDARY OUTCOMES:
Number of patients with emerging or existing macrolide resistance against Mycoplasma genitalium during or after treatment with azithromycin | One month after treatment has started
  Quantitive pcr of chlamydia and Mg is used. All Mg strains are tested for mutant genes.

OTHER OUTCOMES:
Number or rate of patients adherent regarding sampling according to the protocol | One month after starting sampling
  To describe whether the subjects are adherent to the study protocol according to doing the sampling and sending the samples correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Falk, MD PhD, Principal Investigator — Dept of Derm&Venereology Linköping University hospital
Locations (1):
- R&D dept of Local Health Care, Östergötland county council, Linköping, Sweden

REFERENCES:
- [Derived] Falk L, Enger M, Jensen JS. Time to eradication of Mycoplasma genitalium after antibiotic treatment in men and women. J Antimicrob Chemother. 2015 Nov;70(11):3134-40. doi: 10.1093/jac/dkv246. Epub 2015 Aug 17. PMID 26283670